CLINICAL TRIAL: NCT04143516
Title: Clinical Trial Optimizing Tumor Ablation for Liver Metastases: Rapid Tissue Analysis Allowing for Immediate Retreatment; Metabolic Imaging Biomarker Validation; and Predictive Genetic Signatures
Brief Title: Tissue Analysis After Tumor Ablation for Liver Metastases Leading to Immediate Retreatment
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-332
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Liver Metastases
Keywords: Optimizing Tumor Ablation; Rapid Tissue Analysis; Metabolic Imaging Biomarker Validation; Predictive Genetic Signatures; 19-332
MeSH Terms: interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Intervention Model Description: This is a single institution prospective study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients with Liver Metastases (Experimental): The standard of care tumor ablation procedure, post-ablation biopsies and pre- and post-ablation PET scans. If the PET scan is positive (shows areas of cancer in the treated metastases), study participants will undergo additional needle biopsies of the positive areas on the scan. If the biopsies show areas of cancer cells that are still alive, the participants will be immediately retreated with a second ablation procedure.
  Interventions: Diagnostic Test: [18-F]- FDG - PET; Procedure: Tumor ablation (TA); Diagnostic Test: PET/CT Scan

INTERVENTIONS:
Diagnostic Test: [18-F]- FDG - PET — Patients will undergo a limited non-contrast CT and first injection PET to localize the lesion
Procedure: Tumor ablation (TA) — Standard ablation with the intent to create a radius of ablation at least 10 mm larger than the largest lesion diameter in order to achieve a minimum of 5 mm ablation margin around the tumor. Any radiographically-identified and biopsy-confirmed residual tumor will be treated on site with immediate ablation. This repeat ablation is not standard of care but will be performed as described for the initial ablation (in the same procedure session) and follow up will be resumed.
Diagnostic Test: PET/CT Scan — Eligible patients will undergo PET/CT -guided tumor ablation as per standard IR guidelines. All patients will undergo PET/CT again, within approximately 6 weeks (+/- 2 weeks) of tumor ablation to evaluate for CN in the target tumor(s) or any sign of residual tissue enhancement, representing viable residual tumor and incomplete treatment.

SUMMARY:
This study will see whether collecting and analyzing needle biopsy samples from cancer liver metastases after a tumor ablation procedure will be able to identify cancer cells that are still alive. The results of these biopsies could help determine the next treatment for your cancer, but the biopsies could cause side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of liver metastases from various primary tumors
* Confined liver disease or limited extrahepatic disease stable/controlled for at least 4 months (extrahepatic disease amenable to treatment is allowed)
* Lesions of ≤3 cm in maximum diameter
* At least one FDG-avid lesion to be treated***
* INR < 1.5*
* Platelet count ≥ 50,000

Exclusion Criteria:

* Age < 18
* Less than 5 mm distance to a structure (GI or biliary tract), that cannot be protected from ablation injury with technical modifications such as hydro or air dissection
* INR > 1.5 that cannot be corrected with fresh frozen plasma **
* Platelet count of <50,000 that cannot be corrected with transfusion
* More than 3 tumors in the liver
* More than 5 tumors of extrahepatic disease (including mediastinal nodes and pulmonary nodules, abdominal or other lymph nodes, and bone metastasis)
* Presence of any peritoneal Carcinomatosis

  * For patients on Coumadin, general clinical guidelines for IR ablation will be followed.

    * For patients with no FDG-PET avid tumors aim 2 of the protocol will not be assessed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-10-25 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Tumor response | 2 years
  will be measured according to RECIST and PERCIST 1.0. The first CT and PET scan taken after ablation will be considered the new baseline for subsequent comparisons and measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Constantinos Sofocleous, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm